CLINICAL TRIAL: NCT02693080
Title: A Pilot Study of Perfusion CT for Lung Tumors Treated With Stereotactic Ablative Radiation Therapy (SABR)
Brief Title: CT Perfusion Imaging in Predicting Treatment Response in Patients With Non-small Cell Lung Cancer or Lung Metastases Treated With Stereotactic Ablative Radiation Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-31971; NCI-2016-00091 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LUN0072 (Other: OnCore); IRB-31971 (Other: Stanford IRB)
Record Dates: First submitted 2016-01-20; First posted 2016-02-26 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Malignant Lung Neoplasm; Metastatic Malignant Neoplasm in the Lung; Non-Small Cell Lung Carcinoma; Stage IV Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Iopamidol; Iothalamic Acid; Cytidine Triphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Diagnostic (CT perfusion imaging) (Experimental): Patients undergo CT perfusion imaging of the lungs at baseline, within 48 hours of first SABR, and at 2-4 months after completion of SABR. Isovue-200 is used as contrast agent
  Interventions: Device: CAPP-Seq; Drug: Isovue-200; Radiation: Computed Tomography Perfusion Imaging

INTERVENTIONS:
Device: CAPP-Seq — Cancer Personalized Profiling by Deep Sequencing (CAPP-Seq) is an assay which allows quantitative assessment of the levels of circulating-tumor DNA in the blood sample.
  Other Names: Cancer Personalized Profiling by Deep Sequencing
Drug: Isovue-200 — Contrast agent
  Other Names: Lopamidol
Radiation: Computed Tomography Perfusion Imaging
  Other Names: CT Perfusion Imaging

SUMMARY:
This study assesses computed tomography (CT) perfusion imaging in predicting treatment response in patients with non-small cell lung cancer or tumors that have spread from the primary site (place where it started) to the lungs (metastases) treated with stereotactic ablative radiation therapy. CT perfusion imaging is a special type of CT that uses an injected dye in order to see how blood flow through tissues, including lung tissue. CT perfusion imaging of the lungs may help doctors learn whether perfusion characteristics of lung tumors may be predictive of response to treatment and whether lung perfusion characteristics can be used to follow response to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of performing computed tomography (CT) perfusion imaging (CT perfusion imaging) at baseline, within 48 hours post-stereotactic ablative radiation therapy (SABR), and at 2-4 months SABR in patients undergoing SABR for treatment of a lung tumor per standard of care.

SECONDARY OBJECTIVES:

1. To determine the range (variability) of perfusion parameters at baseline, within 48 hours post-SABR, and at 2-4 months post-SABR
2. To assess the change in perfusion parameters at baseline, within 48 hours post-SABR, and at 2-4 months post-SABR
3. To correlate any change in perfusion parameters with circulating-tumor deoxyribonucleic acid (DNA) levels at baseline, within 48 hours post-SABR, and at 2-4 months post-SABR
4. To correlate perfusion parameters with tumor response 1 year post-SABR

OUTLINE:

Patients receive an infusion of Isovue-200 and undergo CT perfusion imaging of the lungs at baseline, within 48 hours of first SABR, and at 2-4 months after completion of SABR. Cancer Personalized Profiling by Deep Sequencing (CAPP-Seq) will be conducted evaluate circulating-tumor DNA levels.

Perfusion parameters will be correlated with tumor control at 1 year post-SABR, with tumor control defined as no evidence of disease seen at the site of SABR by surveillance imaging at 1 year post-SABR.

After completion of treatment, patients are followed up at 2-4 months and then at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing SABR for the treatment of a lung tumor, inclusive of non-small cell lung cancer or lung metastases

Exclusion Criteria:

* Patients who are pregnant or are trying to become pregnant are excluded from this study
* Patients with renal failure, defined as glomerular filtration rate (GFR) < 60 at the time of the radiation treatment-planning (RTP) scan, will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Number of participants able to complete perfusion scan acquisition at the time of treatment-planning | Up to approximately 90 seconds
Number of participants able to complete perfusion scan acquisition within 48 hours of SABR | Within 48 hours post-SABR
Number of participants able to complete perfusion scan acquisition in follow-up up to 4 months after SABR | Up to 4 months post-SABR

SECONDARY OUTCOMES:
The calculated variance of blood flow such that measurable changes can be identified in future studies | Baseline to up to 4 months post-SABR
The calculated variance of blood volume such that measurable changes can be identified in future studies | Baseline to up to 4 months post-SABR
The calculated variance of mean transit time such that measurable changes can be identified in future studies | Baseline to up to 4 months post-SABR
The calculated variance of permeability such that measurable changes can be identified in future studies | Baseline to up to 4 months post-SABR

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Diehn, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

DOCUMENTS (1):
  • Informed Consent Form (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT02693080/ICF_000.pdf